CLINICAL TRIAL: NCT04651244
Title: Diagnostic Imaging of Acute Pyelonephritis - Part of the INDEED Study (Infectious Diseases in Emergency Departments)
Brief Title: Diagnostic Imaging of Acute Pyelonephritis
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Sponsor
Other Study IDs: SHS-ED-11a-2020
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Pyelonephritis Acute
Keywords: Complicated urinary tract infection; Hydronephrosis; Contrast enhanced Ultrasound; Ultrasound; Diagnostic imaging
MeSH Terms: conditions — Hydronephrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected acute pyelonephritis: Patients admitted in the ED with suspected infection, where the initial medical assessment raises suspicion of APN.
  Interventions: Diagnostic Test: MRI; Diagnostic Test: Ultrasound performed by a radiologist; Diagnostic Test: Point of care ultrasound

INTERVENTIONS:
Diagnostic Test: MRI — Gold standard for identifying inflammatory changes in patients with acute pyelonephritis
Diagnostic Test: Ultrasound performed by a radiologist — US performed by a radiologist including standard grayscale evaluation of the kidneys, Doppler US and contrast enhanced US (CEUS).
Diagnostic Test: Point of care ultrasound — Point of care US by a study assistant with basic ultrasound skills and training to access the presence or absence of hydronephrosis. If hydronephrosis is present it will be graded into one of four categories.

SUMMARY:
Acute pyelonephritis is important to recognize and treat quickly. Today the diagnosis is primarily clinical and often challenging. Sometimes acute pyelonephritis is complicated by obstruction leading to hydronephrosis. The aim of this study is to investigate whether ultrasound scanning conducted by a radiologist can diagnose acute pyelonephritis. Also, the investigators will investigate whether health care professionals with basic ultrasound skills can diagnose hydronephrosis by point-of-care ultrasound scanning in patients suspected of acute pyelonephritis.

DETAILED DESCRIPTION:
Acute pyelonephritis (APN) is an acute infection in the upper urinary tract, which quite frequently is seen in emergency departments (ED). Most often, an infection of the bladder ascends to the kidneys causing APN. In rarer cases, APN occurs because of a hematogenous spread of bacteria. It is important to identify and treat APN quickly to prevent progression to sepsis, renal failure and ultimately death. Today, primarily APN diagnosis consists of a clinical identification. This is often supported by unspecific blood and urine tests such as C reactive protein (CRP) and leucocytes and urine dipstick. A positive urine culture verifies the APN diagnosis. This diagnostic process is challenging as frequently symptoms are weak and atypical and there is a waiting period for unspecific diagnostic methods and culture results. Complicating an APN diagnosis is asymptomatic bacteriuria, a confusing condition, common in the elderly. Therefore, the empirical treatment initiated often treats a potentially wide range of infections including APN. Currently, the Danish ED do not use diagnostic imaging to confirm APN. Ultrasound scanning (US) by a radiologist rules out other complicating factors such as obstruction or renal abscess. Further imaging is reserved for complicated cases with no response to the initial treatment. Both Computed Tomography (CT) scanning and Magnetic Resonance Imaging (MRI) can visualize inflammation in the kidneys. Generally, CT is considered the optimal imaging modality in complicated APN cases. The radiation dose-related to a CT must be considered if this imaging technique is to be used as a primary diagnostic tool. MRI appears to be equally or more satisfactory in identifying the inflammatory changes related to APN. However, this investigative tool is more expensive and time-consuming, and often not readily available.

Ultrasound (US) has a lot of advantages in an acute medical setting. It can be utilised at the bedside and is a gentle technique. Conventional grayscale US is not ideal when trying to identify APN. However, more specialized US techniques increase the diagnostic value of US. These techniques include the Doppler US and the contrast-enhanced US (CEUS). Studies suggest that CEUS can identify APN equally to contrast-enhanced CT. Therefore, US has the potential to become relevant in the investigation of patients with a suspected kidney infection in the ED.

This study aims to investigate whether additional diagnostic imaging, in particular US, of patients admitted to the ED with suspected APN will assist in a more reliable diagnosis. Furthermore, it will investigate if point-of-care US of the kidneys by an investigator with basic US skill can assist a more rapid recognition of hydronephrosis in APN patients with complicating obstruction.

The investigators will invite patients admitted with suspected APN to participate in this study, which will include three additional scans. The first is a point of care US of the kidneys by a study assistant to assess the presence or absence of hydronephrosis. The second is a US by a specialist from the Radiology Department using both Doppler US and CEUS. The third scan is a reference standard MRI of the kidneys at the Radiology Department. This will be performed at a similar time (or as close as possible) to the radiologist US. The MRI will be conducted on a 1,5 T MRI scanner and include the following sequences: planning, Dixon, T1 mapping, T2, T2 mapping, apparent diffusion coefficient (ADC) (100, 400, 800), MRI angio (3D VIBE), and Phase Contrast.

These additional imaging findings will be evaluated in relation to the clinical findings.

ELIGIBILITY:
Inclusion Criteria:

* Suspicion of acute pyelonephritis by ED physician
* Suspicion of urinary tract infection by ED physician and systemic affection (e.g. fever, sepsis

Exclusion Criteria:

* Unable to undergo an MRI
* Known allergy to US contrast
* If the attending physician considers that participation will delay a life-saving treatment or patient needs direct transfer to the intensive care unit.
* Admission within the last 14 days
* Verified COVID-19 disease within 14 days before admission
* Pregnant women
* Severe immunodeficiencies: Primary immunodeficiencies and secondary immunodeficiencies (HIV positive CD4 <200, Patients receiving immunosuppressive treatment (ATC L04A), Corticosteroid treatment (>20 mg/day prednisone or equivalent for >14 days within the last 30 days), Chemotherapy within 30 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be included among patients admitted at the ED of three Danish hospitals in the Region of Southern Denmark: the ED in Kolding, Lillebælt Hospital, the ED in Aabenraa, Hospital Sønderjylland, and the ED in Odense, Odense University Hospital.
  A Danish ED corresponds to an acute medical ward. Either a general practitioner or a prehospital emergency medical service refers patients visiting a Danish ED, or patients get admitted because they called the emergency centre telephone number (1-1-2).
Sampling Method: Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Comparison of inflammatory changes in the kidneys on CEUS compared to MRI | Routine descriptions of the scans will be available within about 48 hours from recruitment. Focused descriptions and comparison are conducted within 6 months after investigation.
  Findings on the investigations will be registered on predefined templates. Both kidneys will be described regarding signs of inflammation, where we e.g. look at perfusion on CEUS, and edema or renal lesions on MRI.
  Results of the investigations on the same kidneys are compared in order to access specificity and sensitivity of findings on CEUS compared to MRI.
  The conducting/describing radiologist will be informed of some standardized clinical and paraclinical parameters (e.g. fever, CRP, flank pain, relevant comorbidity), but will be blinded to the results of the other imaging investigations.
Comparison of inflammatory changes in the kidneys on gray scale US and spectral doppler compared to the reference standard MRI | Routine descriptions of the scans will be available within about 48 hours from recruitment. Focused descriptions and comparison is conducted within 6 after investigation.
  Findings on the investigations will be registered on predefined templates. Both kidneys will be described regarding signs of inflammation, where we e.g. look at perfusion and resistance on US, and edema or renal lesions on MRI.
  Results of the investigations on the same kidneys are compared in order to access specificity and sensitivity of findings on US compared to MRI.
  The conducting/describing radiologist will be informed of some standardized clinical and paraclinical parameters (e.g. fever, CRP, flank pain, relevant comorbidity), but will be blinded to the results of the other imaging investigations.
Sensitivity and specificity of point-of-care ultrasound on identifying hydronephrosis compared to MRI | Within 48 hours
  How many of hydronephroses in patients suspected of APN is discovered by point of care US performed by an investigator with basic point of care US skills? MRI of the kidneys conducted maximum 24 hours after the point of care US is used as reference standard.

SECONDARY OUTCOMES:
Proportion of patients with APN and hydronephrosis | Within 12 month
  We use the gold standard investigation, MRI, to evaluate the number of APN patients who also have hydronephrosis.

OTHER OUTCOMES:
Bacteriuria | within 4 hours from admission
  Binary outcome defined by microbiologist on urine culture analysis

CONTACTS AND LOCATIONS:
Overall Officials: Christian Backer Mogensen, Study Chair — Institute for Regional Health Research
Locations (1):
- Hospital of Southern Jutland, Aabenraa, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Claeys KC, Blanco N, Morgan DJ, Leekha S, Sullivan KV. Advances and Challenges in the Diagnosis and Treatment of Urinary Tract Infections: the Need for Diagnostic Stewardship. Curr Infect Dis Rep. 2019 Mar 5;21(4):11. doi: 10.1007/s11908-019-0668-7. PMID 30834993
- [Background] Rathod SB, Kumbhar SS, Nanivadekar A, Aman K. Role of diffusion-weighted MRI in acute pyelonephritis: a prospective study. Acta Radiol. 2015 Feb;56(2):244-9. doi: 10.1177/0284185114520862. Epub 2014 Jan 17. PMID 24443116
- [Background] Cruz J, Figueiredo F, Matos AP, Duarte S, Guerra A, Ramalho M. Infectious and Inflammatory Diseases of the Urinary Tract: Role of MR Imaging. Magn Reson Imaging Clin N Am. 2019 Feb;27(1):59-75. doi: 10.1016/j.mric.2018.09.001. Epub 2018 Oct 29. PMID 30466913
- [Background] Quaia E, Correas JM, Mehta M, Murchison JT, Gennari AG, van Beek EJR. Gray Scale Ultrasound, Color Doppler Ultrasound, and Contrast-Enhanced Ultrasound in Renal Parenchymal Diseases. Ultrasound Q. 2018 Dec;34(4):250-267. doi: 10.1097/RUQ.0000000000000383. PMID 30169495
- [Background] Mitterberger M, Pinggera GM, Colleselli D, Bartsch G, Strasser H, Steppan I, Pallwein L, Friedrich A, Gradl J, Frauscher F. Acute pyelonephritis: comparison of diagnosis with computed tomography and contrast-enhanced ultrasonography. BJU Int. 2008 Feb;101(3):341-4. doi: 10.1111/j.1464-410X.2007.07280.x. Epub 2007 Oct 17. PMID 17941932
- [Background] Kazmierski B, Deurdulian C, Tchelepi H, Grant EG. Applications of contrast-enhanced ultrasound in the kidney. Abdom Radiol (NY). 2018 Apr;43(4):880-898. doi: 10.1007/s00261-017-1307-0. PMID 28856401
- [Derived] Skjot-Arkil H, Heltborg A, Lorentzen MH, Cartuliares MB, Hertz MA, Graumann O, Rosenvinge FS, Petersen ERB, Ostergaard C, Laursen CB, Skovsted TA, Posth S, Chen M, Mogensen CB. Improved diagnostics of infectious diseases in emergency departments: a protocol of a multifaceted multicentre diagnostic study. BMJ Open. 2021 Sep 30;11(9):e049606. doi: 10.1136/bmjopen-2021-049606. PMID 34593497